CLINICAL TRIAL: NCT02080754
Title: Sellick Maneuver Evaluation in Rapid Sequence Induction of General Anesthesia Non Inferiority Trial
Brief Title: Sellick Interest in Rapid Sequence Induction
Acronym: IRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P 120120; 2013-A00624-41 (Other: IDRCB)
Record Dates: First submitted 2014-02-17; First posted 2014-03-06 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-11

CONDITIONS: Rapid Sequence Induction of General Anesthesia; Sellick Maneuver; Acid Aspiration Syndrome; Lung Aspiration; Aspiration Pneumonia
Keywords: Crush induction; Cricoid pressure; Sellick maneuver; Lung aspiration; Aspiration pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham arm (Placebo Comparator): sham sellick maneuver
  Interventions: Other: sham sellick maneuver
- sellick arm (Experimental): effective sellick maneuver
  Interventions: Other: effective sellick maneuver

INTERVENTIONS:
Other: effective sellick maneuver — Sellick maneuver is applied, as originally described by Sellick et al .
  Arms: sellick arm
Other: sham sellick maneuver — The operator who applied the maneuver is the only person who knows the arm inclusion of the patient. Thus, he sets his fingers as described in Sellick arms without exerting pressure on the cricoid cartilage.
  Arms: sham arm

SUMMARY:
Lung aspiration can occur when a rapid sequence induction of anesthesia is performed (emergency and/or presence of at least one risk factor for regurgitation of stomach contents).

The aim of this study is to assess the Sellick maneuver, which is recommended for patient at high risk of aspiration of gastric content during induction of general anesthesia, despite the lack of solid evidence of its efficacy and possible adverse effects The primary outcome of this non inferiority study is the incidence of lung aspiration whether this maneuver is effectively applied or sham.

DETAILED DESCRIPTION:
Introduction:

Lung aspiration is an inherent complication of the loss of protective upper airway reflexes during general anesthesia. Its incidence is low in elective surgery, when preoperative fasting rules have been complied and in absence of risk factors for regurgitation of gastric contents. In emergency conditions, non-compliance with preoperative fasting rules and delayed gastric emptying increase the risk of regurgitation and therefore lung aspiration of gastric contents. In this context, a rapid sequence induction of anaesthesia is recommended to minimize the risk of regurgitation which combines the use of short delay and short duration of action anesthetics agents associated with the application of a Sellick maneuver. The goal of this maneuver is to collapse the esophagus by compressing it between the cricoid cartilage and the fifth cervical vertebra. Because of the low level of evidence supporting the Sellick maneuver in the literature, this maneuver, remains controversial although recommended.

Hypothesis: The aim of this study is to assess the Sellick maneuver during rapid sequence induction in adults (pregnant women excluded) by comparing the incidence of lung aspiration whether this maneuver is applied or sham, in a noninferiority trial.

Primary endpoint: Incidence of lung aspiration

Secondary endpoints: Cormack and Lehane Grade , frequency of difficult intubation, frequency of impossible intubation, effect of releasing the Sellick maneuver on these three criteria, frequency of aspiration pneumonia within 24 hours, frequency of complications due to the Sellick maneuver (esophageal rupture and cricoid cartilage fracture rates) and mortality at day 28 or at hospital discharge.

Methods: This is a multicenter, randomized, double-blind, non-inferiority trial. We compare a group of patients benefiting from a rapid sequence induction without achieving the Sellick maneuver, where the movement is fake (sham group) with a group of patients undergoing a rapid sequence induction with effective execution of this maneuver (Sellick group). The two patient groups differ only by the effective or sham application of the Sellick maneuver .

In both arms, the Sellick maneuver , whether real or fake , can be released at the request of the person performing orotracheal intubation in particular to improve intubating conditions or in case of active vomiting. However, it should be kept in case of need for ventilation facemask.

Number of patients: The number of patients is estimated at 1 750 patients per group and so 3500 patients.

Inclusion criteria: patients older than 18 yr undergoing general anesthesia requiring rapid sequence induction (full stomach or presence of at least one risk factor for regurgitation of stomach content) are eligible.

Exclusion criteria: patients non consenting, pregnancy, contraindication to Sellick maneuver or succinylcholine, patients with predictive signs of bronchopneumonia during the preanesthetic consultation, patients with pulmonary contusion, upper respiratory tract abnormalities, laryngeal trauma, patients requiring an alternative to direct laryngoscopy, patients with troubles of consciousness, use of plastic single used laryngoscopic blade, use of rocuronium as neuromuscular blockade agent.

ELIGIBILITY:
Inclusion criteria :

* Patients older than 18 yr undergoing general anaesthesia requiring rapid sequence induction (full stomach or presence of at least one risk factor for regurgitation of stomach content) are eligible.
* Obtain informed consent from the patient or a close relative/surrogate. Should such a person be absent, the patient will be randomized according to the specifications of emergency consent and the patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.

Exclusion criteria :

* Non consent patients,
* Pregnancy,
* Contraindication to Sellick maneuver
* Contraindication to succinylcholine
* Patients with predictive signs of bronchopneumonia during the preanesthetic consultation ,
* Patients with pulmonary contusion
* Upper respiratory tract abnormalities
* Laryngeal trauma
* Patients requiring an alternative to direct laryngoscopy
* Patients with troubles of consciousness
* Use of plastic single used laryngoscopic blade
* Use of rocuronium as neuromuscular blockade agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3472 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Incidence of lung aspiration | Within 1 hour
  in the operating room presence of gastric fluid on the vocal cords at the orotracheal intubation or in endotracheal suction when performed immediately after intubation

SECONDARY OUTCOMES:
Cormack and Lehane Grade | Within 1 hour
  During orotracheal intubation
Frequency of use of a mask ventilation | Within 1 hour
  In the operating room, if needed, the mask ventilation will be recorded
Number of times the Sellick maneuver should be discontinued | Within 1 hour
  In the operating room, if the person who realize the intubation requires a loosening of the Sellick manoeuver, whether real or feigned (difficult intubation, vomiting)
Effects of releasing the Sellick maneuver on the conditions of tracheal intubation assessed by Cormack and Lehane grade | Within 1 hour
  During orotracheal intubation
Incidence of difficult and impossible intubation | Within 1 hour
  difficult intubation is defined by more than two attempts or the need for an alternative technique. Impossible intubation is defined by the need to awake the patient or perform a tracheotomy or cricothyrotomy rescue.
Incidence of aspiration pneumonia | within the 24 hours
  Aspiration pneumonia is defined by the association of a lung aspiration recorded in the operating room during the induction of anesthesia and the presence of a non-existent preoperative radiological infiltrate
Incidence of oesophageal rupture | day 28
  This complication is extremely rare and clinically very telling. No further review is planned to diagnose it
Incidence of cricoid cartilage fracture | day 28
  This complication is extremely rare and clinically very telling. No further review is planned to diagnose it.
Mortality | day 28
Mortality | Hospital discharge Hospital discharge if anterior at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie Birenbaum, MD, Principal Investigator — APHP
Locations (1):
- Groupe Hospitalier Pitié Salpetriere, Paris, France

REFERENCES:
- [Result] Birenbaum A, Hajage D, Roche S, Ntouba A, Eurin M, Cuvillon P, Rohn A, Compere V, Benhamou D, Biais M, Menut R, Benachi S, Lenfant F, Riou B; IRIS Investigators Group. Effect of Cricoid Pressure Compared With a Sham Procedure in the Rapid Sequence Induction of Anesthesia: The IRIS Randomized Clinical Trial. JAMA Surg. 2019 Jan 1;154(1):9-17. doi: 10.1001/jamasurg.2018.3577. PMID 30347104